CLINICAL TRIAL: NCT05122221
Title: A Phase I Study to Evaluate the Safety, Tolerance and Efficacy of CRTE7A2-01 TCR-T Cell for HPV16 Positive Advanced Cervical, Anal, or Head and Neck Cancers
Brief Title: CRTE7A2-01 TCR-T Cell for HPV-16 Positive Advanced Cervical, Anal, or Head and Neck Cancers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corregene Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRTE7A2-2107C
Record Dates: First submitted 2021-11-05; First posted 2021-11-16 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2021-11

CONDITIONS: Cervical Cancer; Anal Cancer; Head and Neck Cancers
Keywords: 3+3 dose escalation
MeSH Terms: conditions — Uterine Cervical Neoplasms; Anus Neoplasms; Head and Neck Neoplasms | interventions — fludarabine; Cyclophosphamide; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CRTE7A2-01 TCR-T cell therapy (Experimental): Patients will undergo lymphocytapheresis, then treatment with TCR-T cell (at escalating doses) + IL-2
  Interventions: Drug: Fludarabine + Cyclophosphamide; Drug: Interleukin-2; Biological: CRTE7A2-01 TCR-T Cell

INTERVENTIONS:
Drug: Fludarabine + Cyclophosphamide — Fludarabine: 25mg/m²/day×3days Cyclophosphamide: 500mg/m²/day×3 days
Drug: Interleukin-2 — Interleukin-2 20,000,000 IU/time infused within 15 minutes approximately every 8 hours (according to the subject's tolerance, the interval between medications can be extended to 24 hours) for a maximum usage time up to 14 days.
Biological: CRTE7A2-01 TCR-T Cell — On day 0, the TCR-T cells will be administered one time, each bag of cell intravenously within 20 minutes.

SUMMARY:
A single center, open, single arm dose escalation phase I study to evaluate the safety, tolerability, and efficacy of CRTE7A2-01 TCR-T cell for HPV16 positive advanced cervical, anal, or head and neck cancers. The study will determine MTD of CRTE7A2-01 TCR-T cell injection, as well as investigate RP2D.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤65 years.
2. Histologically-confirmed cervical cancer, anal cancer, head and neck cancers with confirmed HPV16 infection and HLA-A*02:01 allele
3. Failure on or intolerance to systemic therapy for unresectable advanced cancer.
4. ECOG performance status of 0-1.
5. Estimated life expectancy ≥ 3 months.
6. Patients must have at least one measurable lesion defined by RECIST 1.1.
7. Female patients of childbearing age must undergo a serum pregnancy test within 7 days prior to study treatment and the results must be negative, and are willing to use a very effective and reliable method of contraception from screening through 6 months after the last dose of study treatment.
8. The patient must be willing to sign the informed consent form and have a good anticipation of compliance with study procedure.

Exclusion Criteria：

1. The proportion of T cell immune-related gene deletion mutations>5%.
2. Patient received any genetically modified T cell therapy.
3. Patient who is being treated with T cell immunosuppressive agent （such as cyclophosphamide, FK506,tripterygium glycosides） or T cell immunoagonist.
4. Patients received chemotherapy, targeted therapy, immunotherapy, or other investigational agents within 2 weeks and received radiotherapy within 4 weeks before apheresis.
5. Patients with any organ dysfuntion as defined below:

   * leukocytes<3.0 x 109/L
   * absolute neutrophil count >1.5 x 109/L
   * hemoglobin<90g/L
   * platelets <100 x 1010/L
   * lymphocytes<0.8 x 109/L
   * percentage of lymphocytes<15%
   * creatinine>1.5×ULN or creatinine clearance <50mL/min
   * total bilirubin>3×ULN; ALT/AST>3×ULN (patients with liver metastasis,>5×ULN)
   * INR>1.5×ULN; APTT>1.5×ULN
   * SpO2≤90%
6. Patients with serious medical conditions, disorders, and / or comorbidities, including, but are not limited to: severe heart disease, cerebrovascular disease, epileptic seizures, uncontrolled diabetes (CTCAE 5.0: FBG ≥ 2 grade), active infection, active digestive tract Ulcer, gastrointestinal bleeding, intestinal obstruction, pulmonary fibrosis, renal failure, respiratory failure.
7. Patient with a severe cardiovascular disease with 6 months before screening, including, but are not limited to, myocardial infarction, severe or unstable angina, coronary or peripheral artery bypass grafting, Heart failure NYHA grade Ⅲ or Ⅳ.
8. Left Ventricular Ejection Fractions (LVEF) <50%.
9. Patient with a known active brain metastases.
10. Patient with a known myelodysplastic syndrome (MDS) or lymphoma.
11. Patient with a known active autoimmune disease, including , but are not limited to, acquired or congenital immunodeficiency disease, allogeneic organ transplantation, autoimmune hepatitis, systemic lupus erythematosus, inflammatory bowel disease.
12. Patient with a known active Hepatitis B or Hepatitis C.
13. Patient with a history of Human Immunodeficiency Virus (HIV) .
14. Patient with a history of syphilis.
15. Pregnant or lactating women.
16. Patient with a known active mental and neurological diseases.
17. The principal investigator judged that it is not suitable to participate in this clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-07-17 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
MTD | 28 days
  Maximum Tolerated Dose
DLT | 28 days
  Dose-limiting toxicity
RP2D | 28 days
  Recommended Phase II Dose
Incidence of treatment related AEs, AEs of special interest and serious adverse events (SAEs). | 2 years
  grade 1-5 (CTCAE)

SECONDARY OUTCOMES:
Objective Response Rate（ORR） | 2 years
  Assessed by RECIST 1.1
Disease Control Rate（DCR） | 2 years
  Assessed by RECIST 1.1
Duration of Response（DOR） | 2 years
  Assessed by RECIST 1.1
Progression-Free Survival（PFS） | 2 years
  Assessed by RECIST 1.1

OTHER OUTCOMES:
Peripheral blood TCR-T cell copy number | 2 years
Negative conversion rate among HPV-16 positive patients detected by tissue biopsy | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No